CLINICAL TRIAL: NCT05542043
Title: Risk Factors for Postpartum Hemorrhage in Patients With Histologically Verified Placenta Accreta
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01047; sp20Ghaemmaghami
Record Dates: First submitted 2022-09-05; First posted 2022-09-15 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Postpartum Hemorrhage (PPH); Placental Dysfunction
Keywords: Placenta Histology; Placenta accreta; Placenta increta; Placenta percreta
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta Accreta | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with normal blood loss (BV < 500 mL)
  Interventions: Other: Data collection
- Women with increased blood loss (BV ≥ 500 mL)
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The data includes anamnestic and clinical data from women whose placental histology reveals a diagnosis of placental dysfunction.
  Maternal data on the following characteristics: age, ethnicity, BMI, pregnancy, parity, number of abortions without curettage, multiple births, previous birth mode.
  Risk factors for placentation disorders (increased maternal age, increased pregnancy and parity, increased BMI, placenta previa, nicotine abuse, multiple births, hypertension, diabetes, infections, bleeding, abortion curettage, hysteroscopy ± cavum curettage, caesarean section, fibroid removal, Asherman' s syndrome, status after IVF, endometritis) and birth mode.
  Data on peripartal and postpartum surgical measures.

SUMMARY:
This retrospective, monocentric study aims to examine risk factors for postpartum hemorrhage in women with histologically verified placenta accreta. Women with histologically verified placenta accreta are divided into two groups: women with normal blood loss (BV < 500 ml) versus women with increased blood loss (BV ≥ 500 ml). The clinical data of pregnant women with histologically verified placental disorders, who gave birth in the Women's Clinic University Hospital Basel (USB) between 1986 and 2019, are compared with each other.

DETAILED DESCRIPTION:
Placental disorders are defined as abnormal implantation of the placenta due to a defect in the basal decidua. Depending on the severity of the incorrect implantation, three different stages can be distinguished (placenta accreta, increta and percreta). Placentation disorders are reported in the literature with an increasing frequency of up to 3%. In the last 10 years, the incidence has increased 10-fold and currently affects 1 to 80 out of 2500 births, depending on the literature. Not every histologically verified placental disorder is associated with postpartum hemorrhage. According to the World Health Organization (WHO), postpartum hemorrhage (PPH) is defined as blood loss ≥ 500 ml within 24 hours after delivery. This retrospective, monocentric study aims to examine risk factors for postpartum hemorrhage in women with histologically verified placenta accreta. Women with histologically verified placenta accreta are divided into two groups: women with normal blood loss (BV < 500 ml) versus women with increased blood loss (BV ≥ 500 ml). The clinical data of pregnant women with histologically verified placental disorders, who gave birth in the Women's Clinic USB between 1986 and 2019, are compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a histologically verified placental disorder who gave birth at the Women's Hospital USB between 1986 and 2019

Exclusion Criteria:

* Existence of a documented refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with histologically verified placental disorder who gave birth in the USB women's clinic between 1986 and 2019.
Sampling Method: Probability Sample
Enrollment: 2348 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Placenta praevia | one time assessment at baseline
  Descriptive analysis: Number of women with Placenta praevia (in women with PPH (blood loss ≥ 500 ml) compared to women with normal blood loss (< 500 ml))
Number of Caesarean sections | one time assessment at baseline
  Descriptive analysis: Number of women with Caesarean section (in women with PPH (blood loss ≥ 500 ml) compared to women with normal blood loss (< 500 ml))
Number of women with obesity | one time assessment at baseline
  Descriptive analysis: Number of pregnant women with obesity (in women with PPH (blood loss ≥ 500 ml) compared to women with normal blood loss (< 500 ml))
Increased maternal age | one time assessment at baseline
  Descriptive analysis: Number of pregnant women with increased maternal age (in women with PPH (blood loss ≥ 500 ml) compared to women with normal blood loss (< 500 ml))

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hoesli, Prof. Dr. med., Principal Investigator — University Hospital Basel, Women's Clinic
Locations (1):
- University Hospital Basel, Women's Clinic, Obstetrics and pregnancy medicine, Basel, Switzerland

REFERENCES:
- [Derived] Ghaem Maghami N, Helfenstein F, Manegold-Brauer G, Amstad G. Risk factors for postpartum haemorrhage in women with histologically verified placenta accreta spectrum disorders: a retrospective single-centre cross-sectional study. BMC Pregnancy Childbirth. 2023 Nov 11;23(1):786. doi: 10.1186/s12884-023-06103-5. PMID 37951863